CLINICAL TRIAL: NCT05301023
Title: Individualized Antibiotic Therapy Versus Standard Care in Children With Febrile Urinary Tract Infection
Brief Title: Individualized Antibiotic Therapy in Children With Acute Uncomplicated Febrile Urinary Tract Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21057310 (UVI RCT)
Record Dates: First submitted 2022-03-11; First posted 2022-03-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Febrile Urinary Tract Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual group (Experimental): In the individual group, the participants receive individualized antibiotic therapy.
  Interventions: Other: Individualized antibiotic therapy
- Standard group (Active Comparator): In the standard group, the participants receive standard antibiotic therapy as defined by the national guideline.
  Interventions: Other: Standard antibiotic therapy

INTERVENTIONS:
Other: Individualized antibiotic therapy — Individualized antibiotic therapy is based on the duration of illness after treatment initiation, as the antibiotic therapy can be stopped three days after the participant has become healthy. The participant is classified as healthy if he/she is afebrile (<38.0 °C), has experienced significant clinical improvement, and have no flank pains or dysuria.
  Arms: Individual group
Other: Standard antibiotic therapy — Standard antibiotic therapy is 10 days of antibiotic therapy regardless of the duration of illness after treatment initiation.
  Arms: Standard group

SUMMARY:
An investigator-initiated, open-label, multi-center, randomized, non-inferiority trial of children aged 3 months to 13 years with acute uncomplicated febrile urinary tract infection. The primary objective is to determine whether individualized antibiotic therapy based on an algorithm (experimental arm) versus standard antibiotic therapy of 10 days (control arm) can reduce the number of days with antibiotic therapy within 28 days after treatment initiation without increasing the risk of recurrent urinary tract infection regardless of the pathogen or death of any cause within 28 days after end of treatment. Children will be randomized 1:1. The medical treatments received are identical in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical suspicion of febrile (≥38 °C) urinary tract infection.
2. Positive urine culture of uropathogenic bacteria obtained by either suprapubic bladder aspiration, sterile intermittent catheterization, or midstream urine.

   1. Suprapubic bladder aspiration: any growth of bacteria.
   2. Sterile intermittent catheterization: monoculture with ≥10^3 cfu/ml.
   3. Midstream urine x 2: Monoculture with the bacteria in both tests with ≥10^4 cfu/ml.
   4. Midstream urine x 2: Monoculture with the bacteria in both tests with ≥10^5 cfu/ml in one test and 10^3 cfu/ml in another test.
   5. Midstream urine x 1 (≥10 years of age): Monoculture with ≥10^5 cfu/ml.
3. 3 months to 13 years of age (corrected age in case of premature birth).
4. Parents fluent in Danish or English.
5. Informed consent both parents.

All children who do not receive any empirical antibiotic therapy but have a positive urine culture (approximately 48 hours after urine sample collection) can be included if fever (≥ 38.0 °C) is present and the child is initiated with relevant antibiotic therapy. ¨

Children can be included regardless of whether intravenous or oral antibiotics were given as empirical therapy.

Exclusion Criteria:

1. Non-Danish civil registration number.
2. Not resident in the Capital Region or Region Zealand in Denmark at primary visit.
3. Previous inclusion in the trial.
4. History of febrile (≥38 °C) urinary tract infection in the last 28 days before the primary visit.
5. Antibiotic treatment in the last two weeks before the primary visit.
6. Three or more episodes with febrile (≥38 °C) urinary tract infection within one year of the primary visit (including the current episode).
7. Previous complicated episode of febrile (≥38 °C) urinary tract infection (e.g., renal abscess or urosepticemia)
8. Non-compliance ≥3 doses of antibiotics during empirical therapy.
9. Elevated creatinine.
10. Prophylactic antibiotic treatment.
11. Known urogenital abnormalities (i.e., obstructing uropathies; vesicoureteral reflux; multicystic dysplasia; renal dysplasia; renal hypoplasia; renal agenesis; duplex kidney; polycystic kidney disease; neurogenic bladder dysfunction; hypospadias).
12. Septic.
13. Positive blood culture (if contamination is not suspected).
14. Immune deficiency.
15. Systemic immunosuppressive therapy.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with recurrent urinary tract infection regardless of the pathogen or death of any cause | within 28 days after end of treatment
Number of days with antibiotic therapy | within 28 days after treatment initiation

SECONDARY OUTCOMES:
Number of days with absence from school or daycare due to illness | within 28 days after randomization
Proportion of participants with recurrent urinary tract infection regardless of the pathogen or death of any cause | within 100 days after end of treatment

OTHER OUTCOMES:
Number of hospital days related to urinary tract infection symptoms | within 28 days after end of treatment
Number of days with a physical or virtual (phone or online) consultation | From date of randomization until the date of treatment stop for the baseline infection, assessed up to 14 days
Proportion of participants with recurrent infection with a bacterium resistant to the antibiotic given for the primary infection | within 100 days after end of treatment
Proportion of participants with a serious adverse event | within 100 days after randomization
  Defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability, or jeopardizes the patient
Proportion of participants with an antibiotic-related non-serious adverse event | within 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Naqash Sethi, MD, Principal Investigator — Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen, Denmark; Ulrikka Nygaard, Ass. prof, Ph.D., Study Chair — Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen, Denmark
Locations (8):
- Denmark (8):
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Copenhagen University Hospital Herlev, Herlev
  - Copenhagen University Hospital Hillerød, Hillerød
  - Copenhagen University Hospital Holbæk, Holbæk
  - Copenhagen University Hospital Hvidovre, Hvidovre
  - Copenhagen University Hospital Nykøbing Falster, Nykøbing Falster
  - Copenhagen University Hospital Roskilde, Roskilde
  - Copenhagen University Hospital Slagelse, Slagelse

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be shared. Individual participant data (IPD) will be shared to facilitate the conduction of systematic reviews with meta-analysis of individual participant data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Primarily for the conduction of individual participant data meta-analysis.

REFERENCES:
- [Derived] Sethi NJ, Carlsen ELM, Tabassum A, Cortes D, Mark Ow S, Schmidt IM, Christensen MM, Kirkedal AK, Kai CM, Bjerre CK, Jensen LH, Antonova M, Sonderkaer S, Rytter MJH, Tordrup G, Zaharov T, Sehested LT, Nygaard U. Efficacy and safety of individualised versus standard 10-day antibiotic treatment in children with febrile urinary tract infection (INDI-UTI): a pragmatic, open-label, multicentre, randomised, controlled, non-inferiority trial in Denmark. Lancet Infect Dis. 2025 Aug;25(8):925-935. doi: 10.1016/S1473-3099(25)00075-1. Epub 2025 Apr 2. PMID 40187361
- [Derived] Sethi N, Carlsen ELM, Schmidt IM, Cortes D, Nygaard U, Sehested LT. Individualised versus standard duration of antibiotic therapy in children with acute uncomplicated febrile urinary tract infection: a study protocol and statistical analysis plan for a multicentre randomised clinical trial. BMJ Open. 2023 Jun 9;13(6):e070888. doi: 10.1136/bmjopen-2022-070888. PMID 37295836